CLINICAL TRIAL: NCT01656486
Title: Utilization of Stereotactic Radiation in Patients With Pancreatic Fistula to Decrease Pancreatic Secretions
Brief Title: Stereotactic Radiation to Decrease Pancreatic Secretions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 07-12-16EM
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2014-02

CONDITIONS: Pancreatic Fistulae
Keywords: Pancreas; Pancreatic fistula; Stereotactic radiation
MeSH Terms: conditions — Pancreatic Fistula | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Radiation (Experimental): Treatment of pancreas with 30 Gy of radiation given in 5 fractions of 6 Gy each with stereotactic radiosurgery.
  Interventions: Radiation: Stereotactic Radiation

INTERVENTIONS:
Radiation: Stereotactic Radiation — Treatment of pancreas with 30 Gy of radiation given in 5 fractions of 6 Gy each with stereotactic radiosurgery that could produce a fibrosis of the pancreas and a decrease in the production of exocrine portion of the gland.

SUMMARY:
Patients that have undergone pre-operative radiation for pancreatic carcinoma, that upon pathologic examination of the normal portion of the pancreatic gland that was in the radiation field showed acute and chronic changes in the pancreatic cells. The hypothesis for utilizing stereotactic radiation on pancreatic fistulae is that the treatment will decrease pancreatic secretions, thus decreasing autodigestion.

DETAILED DESCRIPTION:
Stereotactic radiation for cancer has been utilized to successfully treat the head of the pancreas, which is generally a well-tolerated procedure with minimal complications. Upon further investigation under the microscope, after resection during a complex Whipple operation, it is noted that particularly the exocrine glandular tissue atrophied substantially. Based on this information, the hypothesis for utilizing stereotactic radiation on the remaining pancreas is production of a fibrosis of the pancreas and a decrease in the production of exocrine portion of the gland. The use of stereotactic radiation will be performed on individuals that are non-surgical candidates.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic fistula
* Non-surgical candidate

Exclusion Criteria:

* Surgical candidate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Sindram, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stereotactic Radiation
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Radiation
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (0)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender, Male/Female
  Participants
    Female | 0
    Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Decreased Secretions
Description: Measurement of pancreatic panel, decreased Pancreatic Secretions
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Stereotactic Radiation
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Stereotactic Radiation
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No